CLINICAL TRIAL: NCT04416750
Title: Positioning Imatinib for Pulmonary Arterial Hypertension
Acronym: PIPAH
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Imperial College London (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); Medical Research Council (Other Government); University of Cambridge (Other); University of Sheffield (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRAS ID: 274093; 2020-001157-48 (EudraCT Number); 20HH5896 (Other: Sponsor (Imperial College London)); 20/SC/0240 (Other: Health Research Authority (UK))
Record Dates: First submitted 2020-05-28; First posted 2020-06-04 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Pulmonary Arterial Hypertension; PAH; Imatinib; TKI; Genotype
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Imatinib Mesylate; Therapeutics

STUDY DESIGN:
Intervention Model Description: The highest tolerated dose of Imatinib determined using a Bayesian continual reassessment method. In the first part, 13 patients were recruited sequentially by protocol at a minimum of 4 week intervals. Each patient was administered a dose of imatinib between 100mg and 400mg daily. The selected dose for each patient was based upon the safety and tolerability of doses administered to preceding recruits using a Bayesian continuous reassessment method. The inclusion of patients with implanted monitoring devices allowed us to collect data on an early efficacy marker alongside data on safety and tolerability. With a small extension, we gained further data on the effect of imatinib on cardiopulmonary haemodynamics and activity in PAH patients, covering the full 100mg to 400mg dose range.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Open label; Imatinib tablets administered once daily; Dosage: in the range of 100mg-400mg; Group evaluated: adults with PAH
  Interventions: Drug: Imatinib Mesylate

INTERVENTIONS:
Drug: Imatinib Mesylate — Treatment with Imatinib
  Other Names: Oral treatment

SUMMARY:
Pulmonary Arterial Hypertension (PAH) is a rare condition in which a narrowing of blood vessels carrying blood through the lungs puts an increased work load on the heart; it has to work harder to pump blood through the lungs. While current treatments relieve some of the symptoms, they do not stop or reverse the disease in the affected blood vessels. Imatinib is a medicine licensed for some types of cancers. A published study has shown that imatinib can have beneficial effects on blood flow through the lungs and exercise capacity in patients with PAH, even when added to existing treatments. However, there have been concerns about its safety and tolerability. Imatinib continues to be prescribed occasionally on compassionate grounds, usually when other treatment options have been exhausted, and some patients feel better on the drug. To improve the investigator's understanding, the investigators of this study re-visits the use of Imatinib as a potential treatment for patients with PAH.

DETAILED DESCRIPTION:
What does the study involve?

The study involves treatment of PAH patients with imatinib (study drug) for up to 24 weeks, and clinical assessments and tests to assess the drug's safety and tolerability.

PAH patients will be seen at their local hospital by the PAH clinical research team. Before someone can start study, the study doctor (or clinical study team) will describe the clinical trial in detail. If a potential subject decides to participate, he/she will be asked to sign the informed consent form before any study procedures are done.

Participants will be asked to come to their local hospital for clinical appointments. This includes a screening visit, a baseline visit, three clinical assessments and an end-of-study visit. In between, and at the very end of these, there will be six tele-visits (assessments over the phone). Each clinical appointment will be on a weekday morning or afternoon. No major lifestyle restrictions are required for these appointments.

Participants will undergo clinical examinations and tests to monitor the severity of PAH and the response to the study drug. Clinical procedures include:

* Questions about demographics, medical and medication history
* Physical examination and record of vital signs (blood pressure, temperature, heart and respiratory rate)
* Questionnaire about quality of life,
* Assessments of PAH severity (WHO Functional Class, six-minute walk test, and Borg dyspnoea index)
* Right heart catheterisation to assess response to the drug
* Haematology and clinical chemistry blood tests to ensure safety
* Serum pregnancy test and urine pregnancy tests (if applicable) to exclude pregnancy
* Blood samples to measure the levels of the study drug in the circulation
* Additional blood samples for future research on PAH and/or the mechanism of action of the drug
* Electrocardiogram (ECG), and echocardiogram to assess the size, shape, pumping action and the extent of any damage to the heart
* Brain MRI scan (or CT scan if MR is not indicated/tolerated) to exclude bleeding in the brain

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged between 18-80 years old
2. PAH which is idiopathic; PAH heritable; PAH associated with connective tissue disease; PAH after ≥ 1 year repair of congenital systemic to pulmonary shunt, or PAH associated with anorexigens or other drugs
3. Subjects willing to be genotyped for genes that influence PDGF activity
4. Resting mean pulmonary artery pressure ≥25 mmHg, Pulmonary capillary wedge pressure ≤15 mmHg, PVR >5 wood units, and normal or reduced cardiac output , as measured by right heart catheterisation (RHC) at entry
5. Six-minute walking distance >50m at entry
6. Stable on an unchanged PAH therapeutic regime comprising at least 2 therapies licensed for PAH (any combination of endothelin receptor antagonist, phosphodiesterase inhibitor or prostacyclin analogue) for at least 1 month prior to screening
7. Able to provide written informed consent prior to any study mandated procedures
8. Contraception: Fertile females (women of childbearing potential) are eligible to participate after a negative highly sensitive pregnancy test, if they are taking a highly effective method of contraception during treatment and until the end of relevant systemic exposure. Fertile males who make use of condom and contraception methods during treatment and until the end of relevant systemic exposure in women of childbearing potential -full details are in included in the research protocol-

Exclusion criteria:

1. Unable to provide informed consent and/or are non-fluent speakers of the English language
2. Hypersensitivity to Imatinib or to any of the excipients
3. Clinically-significant renal disease (confirmed by creatinine clearance <30 ml/min per 1.73m2)
4. Clinically-significant liver disease (confirmed by serum transaminases >3 times than upper normal limit)
5. Patients receiving oral and/or parenteral anticoagulants (this does not apply to single antiplatelet therapy)
6. Anaemia confirmed by haemoglobin concentration <10 g/dl
7. History of thrombocytopenia
8. Individuals known to have haemoglobinopathy sickle cell disease, thalassaemia
9. Hospital admission related to PAH or change in PAH therapy within 3 months prior to screening
10. History of left-sided heart disease and/or clinically significant cardiac disease, including but not limited to any of the following:

    1. Aortic or mitral valve disease (stenosis or regurgitation) defined as greater than mild aortic insufficiency, mild aortic stenosis, mild mitral stenosis, moderate mitral regurgitation
    2. Mechanical or bioprosthetic cardiac valve
    3. Pericardial constriction, effusion with tamponade physiology, or abnormal left atrial size.
    4. Restrictive or congestive cardiomyopathy
    5. Left ventricular ejection fraction ≤50% (measured in echocardiogram at screening)
    6. Symptomatic coronary disease
    7. Significant (2+ for regurgitation) valvular disease other than tricuspid or pulmonary regurgitation
    8. Acutely decompensated left heart failure within 1 month of screening
    9. History of untreated obstructive sleep apnoea
11. Evidence of significant lung disease on high-resolution CT (if available) or recent (performed within 12 months) lung function, where FEV1 < 50% predicted and FVC < 70% predicted, and DLCO (or TLCO) < 50% predicted if any CT abnormalities; judged by the Site Physician
12. Patients with a history of uncontrolled systemic hypertension
13. Acute infection (including eye, dental, and skin infections)
14. Chronic inflammatory disease including HIV, and Hepatitis B
15. Women of childbearing potential who are pregnant or breastfeeding (if applicable)
16. Previous intracerebral haemorrhage
17. Patients who have received an Investigational Medicinal Product (IMP) within 5 half-lives of the last dose of the IMP or 1 month (whichever is greater) before the baseline visit

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Identifying the highest tolerated dose | 12 months
  Part 1: Discontinuation of the drug for more than 5 consecutive days due to Grade 2 or above Adverse Events, defined by NCI criteria (version 5.0, 2017) adapted for the study.
Change in pulmonary vascular resistance (PVR) | 24 months
  Part 2: The primary efficacy endpoint is a binary variable. For patients with a baseline pulmonary vascular resistance (PVR) >1000 dynes·s·cm-5, success is defined by an absolute reduction in PVR of ≥300 dynes·s·cm-5 at 24 weeks. For patients with a baseline PVR ≤1000 dynes·s·cm-5, success is a 30% reduction in PVR at 24 weeks.

SECONDARY OUTCOMES:
Change in exercise test | 24 weeks
  Change in six minute walk distance (6MWD) at 24 weeks.
Change in ejection fraction measures | 24 weeks
  Change in right ventricular ejection fraction (RVEF) values, measured in echocardiogram (at screening visit and at 24 weeks).
Change in brain natriuretic peptide (BNP) values | 24 weeks
  Change in plasma BNP (or proNT-BNP) levels from baseline at 24 weeks.
Change in quality of life scores | 24 weeks
  Change in Quality of Life (QoL) scores from baseline at 24 weeks.

OTHER OUTCOMES:
Plasma proteome measures | 24 weeks
  Change in plasma proteome from baseline at 24 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Martin R Wilkins, MD, FRCP, Study Director — Imperial College London
Locations (4):
- United Kingdom (4):
  - Hammersmith Hospital, Imperial College Healthcare NHS Trust, London, Greater London
  - Royal Papworth Hospital, Royal Papworth Hospital NHS Foundation Trust, Cambridge
  - Royal Brompton Hospital, Royal Brompton & Harefield NHS Foundation Trust, London
  - Royal Hallamshire Hospital, Sheffield Teaching Hospitals NHS Foundation, Sheffield